CLINICAL TRIAL: NCT06016621
Title: A Randomised Controlled Trial on the Effectiveness of Improvisational Music Therapy for Autistic Children Aged 7 - 11 [Autism-CHIME Trial].
Brief Title: Autism - Children's Improvisational Music Therapy Evaluation
Acronym: CHIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Simon Baron-Cohen (Other)
Collaborators: Anglia Ruskin University (Other); Musical Universe (Unknown); Rosetrees Trust (Other); Stoneygate Trust (Unknown); Autism Centre of Excellence (Unknown)
Responsible Party: Sponsor-Investigator, Prof Simon Baron-Cohen, Professor Simon Baron-Cohen, University of Cambridge
Organization: University of Cambridge (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRE.2022.077; ETH2223-3184 (Other: Anglia Ruskin University Research Ethics Panel)
Record Dates: First submitted 2023-08-19; First posted 2023-08-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Autism
Keywords: Randomised Controlled Trial; Improvisational music therapy; Autism; Children; Social communication; Social cognition
MeSH Terms: conditions — Autistic Disorder; Communication

STUDY DESIGN:
Intervention Model Description: Assessor-blind, multi-centre, pragmatic, two-arm, randomised controlled trial in which participants will be randomly allocated to either:
  1. Twice-weekly 30 minute-sessions of one to one improvisational music therapy over 12 weeks, in addition to support as usual.
  2. Support as usual control group.
Who Masked: Outcomes Assessor
Masking Description: Research assistants involved in data collection will be blinded to treatment allocation for the entire duration of the study. Success of blinding will be verified by asking assessors if they inadvertently found out about the treatment allocation - instances of unblinding will be recorded using a case report form with details including information on who was unblinded, the source of the unblinding and the reason for the unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Support as usual control Group (No Intervention): Participants allocated to 'support as usual' will receive routine support from their general practitioners (GPs), mental health and education/allied health professionals. Support as usual is defined as normal practice for each school in addition to the usual support from the specialist teaching teams for autism in the area, or any other additional therapies intended to support communication skills or wellbeing for autistic children. They will not receive the individual music therapy intervention or any extra support services from the research team. Any concomitant treatment or therapeutic interventions that participating children might receive will be recorded during assessment sessions before randomisation, and following the primary endpoint, specifying the kind and amount or frequency of intervention.
- Improvisational Music Therapy (Experimental): Participating children randomised to the Improvisational Music Therapy (intervention) Group will receive 30-minute individual music therapy sessions two times per week over a 12-week period. These will be delivered by academically trained Health and Care Professions Council (HCPC)-registered music therapists in the United Kingdom (master's level or equivalent) with clinical experience of working with autistic children. Each child in the intervention arm will receive 24 sessions of music therapy over a 12-week period. A music therapy training manual will be used to guide music therapists.
  Interventions: Behavioral: Improvisational Music Therapy

INTERVENTIONS:
Behavioral: Improvisational Music Therapy — The therapist engages with the child by playing and sharing musical instruments, and/or sings while being attuned to the child's behaviour and expression. Various improvisational techniques are employed to engage the child. There are opportunities for pulse, rhythmic, dynamic or melodic patterns, and timbre to be mirrored, reinforced, or complemented, which allows for moments of synchronization between the therapist and the child, giving the child's musical expressions a pragmatic meaning within this context. The therapist may also gently provoke the child by violating expectations or patterns that have been jointly developed in order to elicit specific social communication behaviours. Further, there are opportunities for the child to develop and enhance social communication skills such as joint attention, sharing affect, reciprocity, shared history, scaffolding, imitation and turn-taking. These have been shown to develop social competency and also resilience.
  Arms: Improvisational Music Therapy

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of individual sessions of improvisational music therapy for autistic children aged 7 - 11.

Researchers will compare the impact of adding improvisational music therapy to usual care alone for autistic children over a 12-week period.

Participants will be randomly assigned to one of the following two conditions: the Improvisational Music Therapy (intervention) Group or the support as usual (control) Group.

The aim is to achieve seven overarching objectives:

1. To determine whether 12 weeks of individual sessions of improvisational music therapy in addition to support as usual is superior to support as usual alone in improving social communication in autistic children.
2. To examine whether 12 weeks of individual sessions of improvisational music therapy in addition to support as usual is superior to support as usual alone in improving communication skills in autistic children.
3. To examine whether 12 weeks of individual sessions of improvisational music therapy in addition to support as usual is superior to support as usual alone in reducing psychosocial problems in autistic children.
4. To examine whether 12 weeks of individual sessions of improvisational music therapy in addition to support as usual is superior to support as usual alone in improving wellbeing of autistic children.
5. To examine whether 12 weeks of individual sessions of improvisational music therapy in addition to support as usual is superior to support as usual alone in improving adaptive functioning in autistic children.
6. To examine whether 12 weeks of individual sessions of improvisational music therapy in addition to support as usual is superior to support as usual alone in improving anxiety in autistic children.
7. To examine whether the therapeutic relationship predicts the development of social, communication and language skills among autistic children.

DETAILED DESCRIPTION:
Co-Chief Investigators Professor Simon Baron-Cohen Dr Carrie Allison Dr David M. Greenberg Dr. Jonathan Pool

Co-Investigators Dr Artur Jaschke

Advisor Emeritus Professor Helen Odell-Miller Dr. Claire Howlin

The Autism-CHIME trial is designed as a rigorous Randomised Controlled Trial (RCT) of individual sessions of improvisational music therapy with autistic children. The trial will be conducted in mainstream and special schools located in Cambridgeshire, Peterborough, London, and the South and East of England. The number of schools involved will depend on the number of eligible children willing to participate, with a minimum of 5-10 children per school.

Enrolled participants will undergo 1:1 block randomisation, to either support as usual plus improvisational music therapy sessions (intervention arm) or support as usual (control arm). Randomisation will occur after the baseline assessments have been completed. Participants will be stratified based on the version of the Brief Observation of Social Communication Change (BOSCC) that they are allocated (primary outcome measure): (1) Minimally Verbal, (2) Phrase Speakers, or (3) Fluent Speakers, so that there are equal numbers in each group, and that the control group and experimental group are balanced.

Data will be collected at different time points during the trial:

The first data collection point (T1) will be collected prior to randomisation (to establish eligibility to participate and assess baseline functioning), and at the primary endpoint T2 (13 weeks after randomisation; end of intervention) and the secondary endpoint T3 will be 39 weeks post-randomisation (i.e. 6 months after the end of music therapy).

The trial will finish after the final follow-up data collection from the participants is completed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7 to 11 years.
* A clinical diagnosis of autism made by a qualified professional according to the International Classification of Diseases (ICD) 10th Revision criteria. Confirmed by a copy of the clinical report detailing the diagnosis (if available) or verified verbally by the child's parents.
* Parents/guardians must give informed consent for their children to be enrolled in the trial.
* Parents/guardians must be willing for the music therapy sessions and BOSCC assessments to be video recorded for monitoring and research purpose
* Participants must be willing to attend two music therapy sessions per week for the duration of the trial.
* Non-verbal children may be included

Exclusion Criteria:

* Received regular individual music therapy in the preceding year as this would be likely to have a strong influence on the course of therapy.
* Severe hearing deficit as this would alter the aim, course, and implementation of therapy.
* Caregivers that are unable to attend for the psychological assessments with their child.
* Caregivers without a basic understanding of English.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Absolute change of the total score of the Brief Observation of Social Communication Change (BOSCC). One of three versions of the BOSCC will be used depending on the child's level of verbal communication. | Baseline and at the end of intervention (13 weeks after randomisation).
  The BOSCC consists of specific items that were developed to identify changes in social-communication behaviours over relatively short periods of time by quantifying subtleties in both the frequency and the quality of specific behaviours. There are three forms of the BOSCC: one for individuals who are minimally verbal (MV), one for those with phrase speech/young fluent speakers (PS/YF up to age 6 - 8) and one for fluent speakers (F1/F2 with two sets of materials, one for children and one for adolescents and adults). Scores are based on the observation of social communicative behaviour during naturalistic interactions between a child and an adult.

SECONDARY OUTCOMES:
Absolute change of the total score of the BOSCC. | Baseline and 39 weeks after randomisation.
  The BOSCC consists of specific items that were developed to identify changes in social-communication behaviours.
Absolute change of the total score of the Children's Communication Checklist-2 to test improvement in communication skills. | Baseline, 13 and 39 weeks after randomisation.
  Measure designed to assess the communication skills of children 4 to 16. It includes two domains: Language (Speech, Syntax, Semantics, Coherence) and Pragmatics (Initiation, Scripted Language, Context, Nonverbal Communication, Social Relations, Interests).
Absolute change of the total score of the Strengths and Difficulties Questionnaire to test improvement in psychosocial difficulties | Baseline, 13 and 39 weeks after randomisation.
  Questionnaire of behavioural and emotional difficulties suitable for children aged 3-16 years old. It addresses different dimensions: emotional problems, conduct problems, hyperactivity/inattention problems, peer problems and prosocial behaviour.
Absolute change of the total score of the Young Child Outcome Rating Scale (YCORS) as a measure of wellbeing. | Baseline, 13 and 39 weeks after randomisation.
  Engaging young children regarding their assessment of how they are doing using child friendly language (faces).
Absolute change of the total score of the Vineland-3 Domain level parent/caregiver form to test improvement in adaptive functioning. | Baseline, 13 and 39 weeks after randomisation.
  Measure of adaptive functioning including Communication domain, Daily living skills domain and Socialization domain.
Absolute change of the total score of the Parent-Rated Anxiety Scale (PRAS) for Youth with Autism Spectrum Disorder (ASD) as a measure of anxiety. | Baseline, 13 and 39 weeks after randomisation.
  The PRAS-ASD is a 25-item, parent-reported measure of anxiety symptoms in youth with ASD (age 5-17 years).
Association between the therapeutic relationship and the development of social, communication and language skills. | Weeks 1 and 12
  The therapeutic relationship will be measured using the Assessment of the Quality of Relationship (AQR), based on video recordings of the first and last of music therapy to evaluate the association between the therapeutic relationship and the development of social, communication and language skills in children allocated to the music therapy intervention.
Absolute change of the total score of the Music Therapy Communication and Social Interaction Scale (MTCSI) (or Music Engagement Scale, MES) based on video recordings. | Weeks 1 and 12.
  Measured based on video recordings of the first and last weeks of music therapy in all of the children allocated to the music therapy intervention) to evaluate communicative and socially interactive responses that are elicited during music therapy sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Pool, PhD, Principal Investigator — Cambridge Institute for Music Therapy Research. Anglia Ruskin University, Cambridge; David M. David M. Greenberg, PhD, Principal Investigator — Musical Universe Inc. USA
Locations (2):
- United Kingdom (2):
  - Anglia Ruskin University, Cambridge
  - Autism Research Centre, Cambridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levitin, D. J. This is your brain on music: The science of a human obsession. vi, 314 (Dutton/Penguin Books, 2006).
- [Background] Savage PE, Loui P, Tarr B, Schachner A, Glowacki L, Mithen S, Fitch WT. Music as a coevolved system for social bonding. Behav Brain Sci. 2020 Aug 20;44:e59. doi: 10.1017/S0140525X20000333. PMID 32814608
- [Background] Sharda M, Tuerk C, Chowdhury R, Jamey K, Foster N, Custo-Blanch M, Tan M, Nadig A, Hyde K. Music improves social communication and auditory-motor connectivity in children with autism. Transl Psychiatry. 2018 Oct 23;8(1):231. doi: 10.1038/s41398-018-0287-3. PMID 30352997
- [Background] American Music Therapy Association (AMTA). https://www.musictherapy.org/.
- [Background] Diagnostic and statistical manual of mental disorders: DSM-5TM, 5th ed. xliv, 947 (American Psychiatric Publishing, Inc., 2013). doi:10.1176/appi.books.9780890425596.
- [Background] Kanner L. Autistic disturbances of affective contact. Acta Paedopsychiatr. 1968;35(4):100-36. No abstract available. PMID 4880460
- [Background] Stegemann T, Geretsegger M, Phan Quoc E, Riedl H, Smetana M. Music Therapy and Other Music-Based Interventions in Pediatric Health Care: An Overview. Medicines (Basel). 2019 Feb 14;6(1):25. doi: 10.3390/medicines6010025. PMID 30769834
- [Background] Lim HA, Draper E. The effects of music therapy incorporated with applied behavior analysis verbal behavior approach for children with autism spectrum disorders. J Music Ther. 2011 Winter;48(4):532-50. doi: 10.1093/jmt/48.4.532. PMID 22506303
- [Background] Lim HA. Effect of "developmental speech and language training through music" on speech production in children with autism spectrum disorders. J Music Ther. 2010 Spring;47(1):2-26. doi: 10.1093/jmt/47.1.2. PMID 20635521
- [Background] Carpente, J. A. Investigating the Effectiveness of a Developmental, Individual Difference, Relationship-Based (DIR) Improvisational Music Therapy Program on Social Communication for Children with Autism Spectrum Disorder. Music Therapy Perspectives 35, 160-174 (2017).
- [Background] Thompson GA, McFerran KS, Gold C. Family-centred music therapy to promote social engagement in young children with severe autism spectrum disorder: a randomized controlled study. Child Care Health Dev. 2014 Nov;40(6):840-52. doi: 10.1111/cch.12121. Epub 2013 Nov 22. PMID 24261547
- [Background] Walworth DD. The use of music therapy within the SCERTS model for children with Autism Spectrum Disorder. J Music Ther. 2007 Spring;44(1):2-22. doi: 10.1093/jmt/44.1.2. PMID 17419661
- [Background] Walworth DD, Register D, Engel JN. Using the SCERTS model assessment tool to identify music therapy goals for clients with autism spectrum disorder. J Music Ther. 2009 Fall;46(3):204-16. doi: 10.1093/jmt/46.3.204. PMID 19757876
- [Background] LaGasse AB. Effects of a music therapy group intervention on enhancing social skills in children with autism. J Music Ther. 2014 Fall;51(3):250-75. doi: 10.1093/jmt/thu012. Epub 2014 Jul 22. PMID 25053766
- [Background] Kim J, Wigram T, Gold C. The effects of improvisational music therapy on joint attention behaviors in autistic children: a randomized controlled study. J Autism Dev Disord. 2008 Oct;38(9):1758-66. doi: 10.1007/s10803-008-0566-6. Epub 2008 Jul 1. PMID 18592368
- [Background] Geretsegger M, Holck U, Carpente JA, Elefant C, Kim J, Gold C. Common Characteristics of Improvisational Approaches in Music Therapy for Children with Autism Spectrum Disorder: Developing Treatment Guidelines. J Music Ther. 2015 Summer;52(2):258-81. doi: 10.1093/jmt/thv005. Epub 2015 May 26. PMID 26019303
- [Background] Howlin C, Rooney B. Cognitive agency in music interventions: Increased perceived control of music predicts increased pain tolerance. Eur J Pain. 2021 Sep;25(8):1712-1722. doi: 10.1002/ejp.1780. Epub 2021 May 6. PMID 33864330
- [Background] Howlin C, Stapleton A, Rooney B. Tune out pain: Agency and active engagement predict decreases in pain intensity after music listening. PLoS One. 2022 Aug 3;17(8):e0271329. doi: 10.1371/journal.pone.0271329. eCollection 2022. PMID 35921262
- [Background] Saarikallio SH, Randall WM, Baltazar M. Music Listening for Supporting Adolescents' Sense of Agency in Daily Life. Front Psychol. 2020 Jan 8;10:2911. doi: 10.3389/fpsyg.2019.02911. eCollection 2019. PMID 32010014
- [Background] Fritz TH, Bowling DL, Contier O, Grant J, Schneider L, Lederer A, Hoer F, Busch E, Villringer A. Musical Agency during Physical Exercise Decreases Pain. Front Psychol. 2018 Jan 17;8:2312. doi: 10.3389/fpsyg.2017.02312. eCollection 2017. PMID 29387030
- [Background] Geretsegger M, Elefant C, Mossler KA, Gold C. Music therapy for people with autism spectrum disorder. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD004381. doi: 10.1002/14651858.CD004381.pub3. PMID 24936966
- [Background] Gold C, Wigram T, Elefant C. Music therapy for autistic spectrum disorder. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004381. doi: 10.1002/14651858.CD004381.pub2. PMID 16625601
- [Background] Whipple J. Music in intervention for children and adolescents with autism: a meta-analysis. J Music Ther. 2004 Summer;41(2):90-106. doi: 10.1093/jmt/41.2.90. PMID 15307805
- [Background] Ozdemir E, Norton A, Schlaug G. Shared and distinct neural correlates of singing and speaking. Neuroimage. 2006 Nov 1;33(2):628-35. doi: 10.1016/j.neuroimage.2006.07.013. Epub 2006 Sep 7. PMID 16956772
- [Background] Nilsson U. Soothing music can increase oxytocin levels during bed rest after open-heart surgery: a randomised control trial. J Clin Nurs. 2009 Aug;18(15):2153-61. doi: 10.1111/j.1365-2702.2008.02718.x. PMID 19583647
- [Background] Ooishi Y, Mukai H, Watanabe K, Kawato S, Kashino M. Increase in salivary oxytocin and decrease in salivary cortisol after listening to relaxing slow-tempo and exciting fast-tempo music. PLoS One. 2017 Dec 6;12(12):e0189075. doi: 10.1371/journal.pone.0189075. eCollection 2017. PMID 29211795
- [Background] Keeler JR, Roth EA, Neuser BL, Spitsbergen JM, Waters DJ, Vianney JM. The neurochemistry and social flow of singing: bonding and oxytocin. Front Hum Neurosci. 2015 Sep 23;9:518. doi: 10.3389/fnhum.2015.00518. eCollection 2015. PMID 26441614
- [Background] Schladt TM, Nordmann GC, Emilius R, Kudielka BM, de Jong TR, Neumann ID. Choir versus Solo Singing: Effects on Mood, and Salivary Oxytocin and Cortisol Concentrations. Front Hum Neurosci. 2017 Sep 14;11:430. doi: 10.3389/fnhum.2017.00430. eCollection 2017. PMID 28959197
- [Background] Feldman R. Sensitive periods in human social development: New insights from research on oxytocin, synchrony, and high-risk parenting. Dev Psychopathol. 2015 May;27(2):369-95. doi: 10.1017/S0954579415000048. PMID 25997760
- [Background] Shamay-Tsoory SG, Saporta N, Marton-Alper IZ, Gvirts HZ. Herding Brains: A Core Neural Mechanism for Social Alignment. Trends Cogn Sci. 2019 Mar;23(3):174-186. doi: 10.1016/j.tics.2019.01.002. Epub 2019 Jan 21. PMID 30679099
- [Background] Gold BP, Mas-Herrero E, Zeighami Y, Benovoy M, Dagher A, Zatorre RJ. Musical reward prediction errors engage the nucleus accumbens and motivate learning. Proc Natl Acad Sci U S A. 2019 Feb 19;116(8):3310-3315. doi: 10.1073/pnas.1809855116. Epub 2019 Feb 6. PMID 30728301
- [Background] Bieleninik L, Geretsegger M, Mossler K, Assmus J, Thompson G, Gattino G, Elefant C, Gottfried T, Igliozzi R, Muratori F, Suvini F, Kim J, Crawford MJ, Odell-Miller H, Oldfield A, Casey O, Finnemann J, Carpente J, Park AL, Grossi E, Gold C; TIME-A Study Team. Effects of Improvisational Music Therapy vs Enhanced Standard Care on Symptom Severity Among Children With Autism Spectrum Disorder: The TIME-A Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):525-535. doi: 10.1001/jama.2017.9478. PMID 28787504
- [Background] Lord C, Risi S, Lambrecht L, Cook EH Jr, Leventhal BL, DiLavore PC, Pickles A, Rutter M. The autism diagnostic observation schedule-generic: a standard measure of social and communication deficits associated with the spectrum of autism. J Autism Dev Disord. 2000 Jun;30(3):205-23. PMID 11055457
- [Background] Broder-Fingert S, Feinberg E, Silverstein M. Music Therapy for Children With Autism Spectrum Disorder. JAMA. 2017 Aug 8;318(6):523-524. doi: 10.1001/jama.2017.9477. No abstract available. PMID 28787492
- [Background] Mossler K, Gold C, Assmus J, Schumacher K, Calvet C, Reimer S, Iversen G, Schmid W. The Therapeutic Relationship as Predictor of Change in Music Therapy with Young Children with Autism Spectrum Disorder. J Autism Dev Disord. 2019 Jul;49(7):2795-2809. doi: 10.1007/s10803-017-3306-y. PMID 28936692
- [Background] Rabeyron T, Robledo Del Canto JP, Carasco E, Bisson V, Bodeau N, Vrait FX, Berna F, Bonnot O. A randomized controlled trial of 25 sessions comparing music therapy and music listening for children with autism spectrum disorder. Psychiatry Res. 2020 Nov;293:113377. doi: 10.1016/j.psychres.2020.113377. Epub 2020 Aug 8. PMID 32798927
- [Background] Roche L, Adams D, Clark M. Research priorities of the autism community: A systematic review of key stakeholder perspectives. Autism. 2021 Feb;25(2):336-348. doi: 10.1177/1362361320967790. Epub 2020 Nov 3. PMID 33143455
- [Background] Geretsegger M, Fusar-Poli L, Elefant C, Mossler KA, Vitale G, Gold C. Music therapy for autistic people. Cochrane Database Syst Rev. 2022 May 9;5(5):CD004381. doi: 10.1002/14651858.CD004381.pub4. PMID 35532041
- [Background] Grzadzinski R, Carr T, Colombi C, McGuire K, Dufek S, Pickles A, Lord C. Measuring Changes in Social Communication Behaviors: Preliminary Development of the Brief Observation of Social Communication Change (BOSCC). J Autism Dev Disord. 2016 Jul;46(7):2464-79. doi: 10.1007/s10803-016-2782-9. PMID 27062034
- [Background] Norbury CF, Nash M, Baird G, Bishop D. Using a parental checklist to identify diagnostic groups in children with communication impairment: a validation of the Children's Communication Checklist--2. Int J Lang Commun Disord. 2004 Jul-Sep;39(3):345-64. doi: 10.1080/13682820410001654883. PMID 15204445
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Guerrero, N. et al. Music Therapy Communication and Social Interaction Scale - Group. (2014).
- [Background] Auyeung B, Baron-Cohen S, Wheelwright S, Allison C. The Autism Spectrum Quotient: Children's Version (AQ-Child). J Autism Dev Disord. 2008 Aug;38(7):1230-40. doi: 10.1007/s10803-007-0504-z. Epub 2007 Dec 7. PMID 18064550
- [Background] Sigman M, Ruskin E, Arbeile S, Corona R, Dissanayake C, Espinosa M, Kim N, Lopez A, Zierhut C. Continuity and change in the social competence of children with autism, Down syndrome, and developmental delays. Monogr Soc Res Child Dev. 1999;64(1):1-114. doi: 10.1111/1540-5834.00002. PMID 10412222
- [Background] Blauth, L. Music therapy and parent counselling to enhance resilience in young children with autism spectrum disorder: a mixed methods study. (Anglia Ruskin University, 2019).
- [Background] Sharda M, Silani G, Specht K, Tillmann J, Nater U, Gold C. Music therapy for children with autism: investigating social behaviour through music. Lancet Child Adolesc Health. 2019 Nov;3(11):759-761. doi: 10.1016/S2352-4642(19)30265-2. Epub 2019 Sep 4. No abstract available. PMID 31494080
- [Background] Green J, Charman T, McConachie H, Aldred C, Slonims V, Howlin P, Le Couteur A, Leadbitter K, Hudry K, Byford S, Barrett B, Temple K, Macdonald W, Pickles A; PACT Consortium. Parent-mediated communication-focused treatment in children with autism (PACT): a randomised controlled trial. Lancet. 2010 Jun 19;375(9732):2152-60. doi: 10.1016/S0140-6736(10)60587-9. Epub 2010 May 20. PMID 20494434
- [Background] Kasari C, Gulsrud A, Paparella T, Hellemann G, Berry K. Randomized comparative efficacy study of parent-mediated interventions for toddlers with autism. J Consult Clin Psychol. 2015 Jun;83(3):554-63. doi: 10.1037/a0039080. Epub 2015 Mar 30. PMID 25822242
- [Background] Porter S, McConnell T, McLaughlin K, Lynn F, Cardwell C, Braiden HJ, Boylan J, Holmes V; Music in Mind Study Group. Music therapy for children and adolescents with behavioural and emotional problems: a randomised controlled trial. J Child Psychol Psychiatry. 2017 May;58(5):586-594. doi: 10.1111/jcpp.12656. Epub 2016 Oct 27. PMID 27786359
- [Background] Bharathi, G., Venugopal, A. & Vellingiri, B. Music therapy as a therapeutic tool in improving the social skills of autistic children. Egypt J Neurol Psychiatry Neurosurg 55, 44 (2019).
- [Background] Gattino, G. S., Riesgo, R. D. S., Longo, D., Leite, J. C. L. & Faccini, L. S. Effects of relational music therapy on communication of children with autism: a randomized controlled study. Nordic Journal of Music Therapy 20, 142-154 (2011).
- [Background] Gupta SK. Intention-to-treat concept: A review. Perspect Clin Res. 2011 Jul;2(3):109-12. doi: 10.4103/2229-3485.83221. PMID 21897887
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822
- [Derived] Jaschke AC, Howlin C, Pool J, Greenberg YD, Atkinson R, Kovalova A, Merriam E, Pallas-Ferrer I, Williams S, Moore C, Hayden K, Allison C, Odell-Miller H, Baron-Cohen S. Study protocol of a randomized control trial on the effectiveness of improvisational music therapy for autistic children. BMC Psychiatry. 2024 Sep 27;24(1):637. doi: 10.1186/s12888-024-06086-3. PMID 39334042

DOCUMENTS (1):
  • Study Protocol (2023-09-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT06016621/Prot_000.pdf